CLINICAL TRIAL: NCT00843739
Title: Expiratory Muscle Training in Patients With Parkinson's Disease
Acronym: EMST
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HD046903-01A112; HD046903-01A112
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Last update posted 2011-09-20 (Estimated); Status verified 2009-02

CONDITIONS: Parkinson's Disease
Keywords: Breathing; Cough; Speech; Swallow; Parkinson's disease
MeSH Terms: conditions — Parkinson Disease; Respiratory Aspiration; Cough; Speech

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- EMST (Experimental): Four week device driven strength training program
  Interventions: Device: EMST - Active Treatment
- sham (Sham Comparator): Four week sham device driven training program
  Interventions: Device: sham EMST
- Control (No Intervention): Four weeks of no intervention

INTERVENTIONS:
Device: EMST - Active Treatment — Hand held device used for strengthening expiratory muscles
  Other Names: Respiratory Muscle Strength Training
  Arms: EMST
Device: sham EMST — Four week sham device training program
  Arms: sham

SUMMARY:
Respiratory difficulty is one of the primary factors leading to death in patients with Idiopathic Parkinson's Disease (IPD). The progressive degeneration of a family of segregated motor and non-motor circuits in the brain results in motor and non-motor dysfunction. Breathing and swallowing are well known to be affected in IPD, and attention to these functions is fitting since most patients eventually experience morbidity and even mortality as a result of this dysfunction. Patients with IPD typically become sedentary and lose endurance, maximal fitness levels and overall pulmonary function. Much of the research focus has been on the motor symptoms of IPD (tremor, rigidity, bradykinesia) yet the pulmonary complications are perhaps ultimately the most important disability. The inability to generate adequate respiratory pressure is responsible for reduced cough magnitudes and cough response times. Cough is critical for the clearance of foreign materials in the airway helping to reduce infiltration of bacteria and subsequent respiratory infection. With reduced cough function an increased risk for pulmonary disease due to a reduced ability to protect the airways occurs. Moreover, the recognized debilitating disruptions to voice and speech characteristics that limit communication, care taking, employment opportunities and social interactions are also a result of poor respiratory function. There are a number of promising outcomes from an expiratory strength-training program. By increasing expiratory muscle strength and expiratory pressure generation, effective breathing, clearance of the airway, production of a louder and clearer voice as well as improved swallowing can occur. These explicit outcomes are predicted based on our experience with the use of an innovative device-driven, home-based expiratory strength training program focused on the expiratory muscles of respiration.

The aims of this study are to: 1) Investigate the activity of expiratory muscle strength training (EMT) in patients with idiopathic Parkinson's disease (IPD), 2) Determine the effect of increased expiratory force generation on breathing, cough magnitude, speech production, and swallowing, 3) Determine the effect of increased expiratory force generation on the patient's perception of speech change, 4) Determine the effect of Dopamine-replacement therapy (Parkinson's medications) on breathing, coughing, speaking, and swallowing measures.

ELIGIBILITY:
Inclusion Criteria:

* Adults between the age of 35 and 85 years.
* Diagnosis of Idiopathic Parkinson's Disease (either tremor-predominant or rigid- predominant) by their neurologist.
* Disability level of II, III, or IV (Hoehn & Yahr, 1976) as indicated in their most recent neurological evaluation.
* Forced Expiratory Volumes (FEV1) and forced vital capacity (FVC) within normative range for age and sex determined by a pulmonary function screening.
* Persons who are able to maintain their current level of physical activity (including both aerobic exercise and weightlifting) throughout the entire training period.

  *Subjects will be asked to report any significant changes in their level of activity throughout their participation in the study in regards to intensity and frequency of exercise (i.e. a sedentary person begins exercising three to four days per week).
* Completion of the informed consent to participate in the study.

Exclusion Criteria:

* Other neurological disorders
* Positive history of any of the following conditions:

  * Gastrointestinal disease
  * Gastro-esophageal surgery
  * Head or neck cancer
  * History of breathing disorders or diseases (e.g., Asthma, chronic obstructive pulmonary disease (COPD)).
  * Untreated hypertension
  * Heart disease
* History of smoking in the last five years
* Failing the screening test of pulmonary functions (e.g., FEV1/FVC < 75%)
* Difficulty in complying with the training protocol due to neuropsychological dysfunction (e.g., severe depression).
* Other illness that would prevent patient from completing the protocol.

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2004-01; Primary Completion 2007-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Maximum Expiratory Pressure | Four weeks

SECONDARY OUTCOMES:
Penetration-Aspiration Score | Four weeks
Peak Expiratory Flow Rate | Four weeks
Laryngeal Compression Duration | Four weeks
Speech timing | Four weeks

CONTACTS AND LOCATIONS:
Overall Officials: Christine M Sapienza, Ph.D., Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Background] Wheeler-Hegland KM, Rosenbek JC, Sapienza CM. Submental sEMG and hyoid movement during Mendelsohn maneuver, effortful swallow, and expiratory muscle strength training. J Speech Lang Hear Res. 2008 Oct;51(5):1072-87. doi: 10.1044/1092-4388(2008/07-0016). Epub 2008 Aug 26. PMID 18728114
- [Background] Kim J, Davenport P, Sapienza C. Effect of expiratory muscle strength training on elderly cough function. Arch Gerontol Geriatr. 2009 May-Jun;48(3):361-6. doi: 10.1016/j.archger.2008.03.006. Epub 2008 May 23. PMID 18457885
- [Background] Chiara T, Martin D, Sapienza C. Expiratory muscle strength training: speech production outcomes in patients with multiple sclerosis. Neurorehabil Neural Repair. 2007 May-Jun;21(3):239-49. doi: 10.1177/1545968306294737. Epub 2007 Mar 9. PMID 17351085
- [Background] Wheeler KM, Chiara T, Sapienza CM. Surface electromyographic activity of the submental muscles during swallow and expiratory pressure threshold training tasks. Dysphagia. 2007 Apr;22(2):108-16. doi: 10.1007/s00455-006-9061-4. Epub 2007 Feb 10. PMID 17294298
- [Background] Baker S, Davenport P, Sapienza C. Examination of strength training and detraining effects in expiratory muscles. J Speech Lang Hear Res. 2005 Dec;48(6):1325-33. doi: 10.1044/1092-4388(2005/092). PMID 16478374
- [Background] Saleem AF, Sapienza CM, Okun MS. Respiratory muscle strength training: treatment and response duration in a patient with early idiopathic Parkinson's disease. NeuroRehabilitation. 2005;20(4):323-33. PMID 16403998
- [Result] Pitts T, Bolser D, Rosenbek J, Troche M, Okun MS, Sapienza C. Impact of expiratory muscle strength training on voluntary cough and swallow function in Parkinson disease. Chest. 2009 May;135(5):1301-1308. doi: 10.1378/chest.08-1389. Epub 2008 Nov 24. PMID 19029430
- See also: Movement Disorders Center - Univ of Florida — http://mdc.mbi.ufl.edu